CLINICAL TRIAL: NCT00041626
Title: Effectiveness and Safety of INGN 201 in Combination With Chemotherapy Versus Chemotherapy Alone
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Introgen Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T302; NCT00040716 (obsolete NCT alias)
Record Dates: First submitted 2002-07-11; First posted 2002-07-12 (Estimated); Last update posted 2007-09-11 (Estimated); Status verified 2007-09

CONDITIONS: Carcinoma, Squamous Cell
Keywords: Recurrent Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck | interventions — advexin

INTERVENTIONS:
Genetic: INGN 201

SUMMARY:
There is a need for more treatment options for patients with recurrent squamous cell cancer of the head and neck (SCCHN). These tumors usually have a variety of genetic defects that include disruption of the p53 pathway, a pathway that would ordinarily work to prevent the development of tumors. In this study the transfer of the p53 gene to tumor cells using a modified adenovirus (INGN 201) in combination with chemotherapy (cisplatin and fluorouracil) will be compared to chemotherapy with cisplatin and fluorouracil in patients who have failed surgery and radiotherapy.

ELIGIBILITY:
* 18 years or older
* Must have had radiation treatment
* Eligible for chemotherapy
* Not eligible for surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin Menander, MD, Study Director; Julie L Sicam, MT (ASCP) MSHS, Study Chair
Locations (8):
- United States (8):
  - University of Arkansas, Little Rock, Arkansas
  - Unversity of Colorado Cancer Center, Aurora, Colorado
  - University of Miami Hospital and Sylvester Comprehensive Cancer Center, Miami, Florida
  - Norton Healthcare Pavilion, Louisville, Kentucky
  - Center Center of GBMC, Baltimore, Maryland
  - WJB Dorn VA Medical Center, Columbia, South Carolina
  - Mary Crowley Medical Research Center, Dallas, Texas
  - University of Texas, MD Andersen Cancer Center, Houston, Texas